CLINICAL TRIAL: NCT01514955
Title: An Initial Feasibility Study to Integrate High-precision, Image Guided, Radiotherapy(MRI Based Brachytherapy and CT/MRI Fused Dynamic IMRT Planning) in the Treatment Planning of 10 Patients With Locally Advanced Carcinoma of the Cervix
Brief Title: An Initial Feasibility Study to Integrate MRI Based Brachytherapy and CT/MR Fused INRT in Treatment of Advance Cervical Cancer
Acronym: IMRT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: IMRT / 25027; ACRI PILOT GRANT
Record Dates: First submitted 2011-12-08; First posted 2012-01-23 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-01

CONDITIONS: Integrated MRI Based RT as Standard of Care; Locally Advanced Cervical Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Gold seeds insertion to detect movements at pelvis
Radiation: Image guided MRI based RT (IMRT+Brachytherapy)

SUMMARY:
Main cause of mortality in cervix cancer is local relapse in the pelvis. Since distant metastasis is quiet rare, increasing local control in the pelvis can directly translate into improvement in survival. Obstacles in front of this approach is the dose limitation to normal organs located in the pelvis adjacent to the tumor. 3-D MRI based EBRT and Brachytherapy will grant safe delivery of more conformal higher doses of radiation to the tumor and allowing sparing of the normal structures.

DETAILED DESCRIPTION:
A total of 10 patients with a diagnosis of locally advanced cervical carcinoma will be enrolled. After diagnosis and written informed consent, patients will undergo investigations prior to treatment planning, including CT imaging as per standard of care. In addition, patients will have an MRI of the pelvis + PET scan + EUA and gold seeds insertion to verify pelvic organs movement and EB-IMRT with daily cone beam CT. Brachytherapy treatment planning will be based on MRI imaging with the applicator in situ.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the uterine cervix considered suitable for curative treatment with definitive radio-chemo-therapy including MRI guided BT. (stage IB2 bulky disease-stage IVa)
* Staging according to FIGO and TNM guidelines
* Positive biopsy showing squamous cell carcinoma, adenocarcinoma or adeno-squamous cell carcinoma of the uterine cervix
* No pelvic nodes > 2cm
* MRI of pelvis at diagnosis
* MRI of the retroperitoneal space and abdomen at diagnosis
* MRI with applicator in place at time of BT
* Age 18-70 years
* Patient informed consent

Exclusion Criteria:

* Pelvic nodes > 2cm
* Previous pelvic or abdominal radiotherapy
* Previous total or partial hysterectomy
* Combination of preoperative radiotherapy with surgery
* Patients receiving neo-adjuvant chemotherapy
* Patients receiving BT only
* Contraindications to MRI

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Feasibility parameters | One year

SECONDARY OUTCOMES:
Response rate, acute and late toxicity, local control rate, survival | Five years
Dosimetric comparison between 2D and 3D Brachytherapy treatment planning